CLINICAL TRIAL: NCT07277569
Title: Nail Plate Construct in Proximal Femoral Fractures With Lateral Wall Deficiency in Skeletally Mature Patients: A Case Series Study.
Brief Title: Combined Nail and Plate Fixation in Proximal Femoral Fractures With Lateral Wall Deficiency
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelraoof Ali Mohamed Ali Morsy, residant doctor at Assiut university hospital, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUN-Ortho-NailPlate-2025
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Femoral Fractures
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nail plate construct (Active Comparator): Combined intramedullary nail and lateral plate fixation for proximal femoral fractures with lateral wall deficiency. The construct includes a proximal femoral nail (PFN) augmented by a dynamic compression plate (DCP) to enhance stability and maintain reduction.
  Interventions: Procedure: Proximal femoral nail with lateral plate augmentation

INTERVENTIONS:
Procedure: Proximal femoral nail with lateral plate augmentation — Surgical fixation using a proximal femoral nail (PFN) augmented with a dynamic compression plate (DCP). Standard lateral approach; fracture reduction under fluoroscopy; temporary K-wires; plate applied to maintain reduction; PFN inserted and locked; layered closure over suction drain.

SUMMARY:
Proximal femoral fractures are a major cause of hospitalization and disability worldwide (1). They are commonly seen among elderly patients after low-energy trauma and in younger adults after high-energy injuries and represent a major challenge in orthopaedic management (2) (3).

These fractures pose unique biomechanical challenges because of axial compression, bending forces and the strong muscle pull that leads to flexion, abduction and external rotation of the proximal fragment (4). Operative management aims to restore anatomical alignment and length to allow early mobilization and weight bearing (5).

Intramedullary devices are widely considered the preferred option for fixation of intertrochanteric fractures, including both stable and unstable types. Their biomechanical advantages include a shorter lever arm, load sharing properties, reduced bending forces, prevention of proximal fragment lateral migration, nearing to the weight-bearing axis, supporting the medial calcar, and allowance for controlled impaction. Clinically, intramedullary nails are also associated with shorter operative time, less soft tissue dissection, reduced blood loss, and earlier mobilization, leading to improved functional outcomes (6-10).

The integrity of the lateral trochanteric wall plays a crucial role in construct stability by serving as a lateral buttress. Loss of this support results in uncontrolled collapse, medialization of the femoral shaft, excessive varus deformity, and limb shortening (11-12). In a cadaveric investigation, Nie et al. (13) reported that the proximal femoral nail provides adequate support to the medial wall but fails to sufficiently stabilize the lateral wall. Furthermore, clinical evidence has shown that approximately 22% of patients with lateral wall disruption required re-operation due to unsatisfactory initial fixation (14).

To address these challenges, recent studies have proposed combined fixation using an intramedullary nail augmented with a lateral plate, aiming to enhance stability, prevent varus collapse, and improve clinical outcomes in complex proximal femoral fractures (15).

However, evidence supporting this combined approach remains limited, with most available studies being small in scale and heterogeneous. Therefore, reporting outcomes from a case series may provide valuable insights into the feasibility, safety, and effectiveness of combined nail-plate fixation, and may serve as a foundation for future comparative studies.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients
* AO trochanteric fractures 31A2 or 31A3 with lateral wall thickness > 20.5 mm on pre-operative radiographs
* Injury Severity Score (ISS) ≤ 17

Exclusion Criteria:

* Open fractures (Gustilo-Anderson type III)
* Delayed presentation > 3 weeks
* Uncontrolled comorbidities (e.g., uncontrolled diabetes or hypertension; cardiac, renal, hepatic, or respiratory failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic assessment of fracture alignment | 2 weeks, 3 months, and 6 months postoperatively
  Radiographic assessment of fracture alignment and implant position on AP and lateral long-film femur radiographs at 2 weeks, 3 months, and 6 months postoperatively. CT will be performed at 6 months if indicated.

SECONDARY OUTCOMES:
Time to union | Up to 6 months
  Months from surgery to radiographic union on serial imaging.
Implant failure | Up to 6 months
  Any mechanical failure unplanned return to OR.
Complications | Intraoperative to 6 months
  Surgical and medical adverse events recorded prospectively.

OTHER OUTCOMES:
Harris Hip Score (HHS) | 6 weeks, 3 months, 6 months
  The Harris Hip Score is a clinician-reported outcome assessing hip pain and function. Scores range from 0 to 100, with higher scores indicating better hip function.
Visual Analog Scale (VAS) for pain | 6 weeks, 3 months, 6 months
  Pain intensity measured using the Visual Analog Scale. Scores range from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain.
Short Form-36 (SF-36) | 6 weeks, 3 months, 6 months
  The Short Form-36 assesses health-related quality of life across eight domains. Each domain is scored from 0 to 100, with higher scores indicating better health-related quality of life.

IPD SHARING:
Plan to Share IPD: No